CLINICAL TRIAL: NCT03434639
Title: Non-invasive Transcutaneous Spectroscopy for the Assessment of Gut Permeability
Brief Title: Fluorescence Spectroscopy for Gut Permeability Assessment
Acronym: GutPerm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Alexander Thompson, Dr Alex Thompson (Imperial College Research Fellow), Imperial College London
Other Study IDs: 18SM4374
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Development and Validation of Gut Permeability Sensor; Permeability; Increased; Celiac Disease; Inflammatory Bowel Diseases; Liver Diseases; HIV/AIDS
Keywords: Gut permeability; Fluorescence; Spectroscopy; Wearable sensor; Leaky gut
MeSH Terms: conditions — Celiac Disease; Inflammatory Bowel Diseases; Liver Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of urine, blood, stool and/or intestinal tissue will be collected from certain participants. Where consent allows, remaining samples will be retained in the Imperial College BioBank after completion of the study for a total of 10 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1 - Ophthalmology patients: Ophthalmology patients who are receiving an intravenous dose of either fluorescein or indocyanine green (ICG) as part of their routine ophthalmic care (e.g. as part of a fluorescence angiography examination) will be recruited to the first stage of this study. These patients will take part in preliminary studies aimed at determining whether it is possible to detect fluorescein and ICG in the blood using transcutaneous fluorescence measurements.
  Interventions: Diagnostic Test: Spectroscopic gut permeability test
- 2a - Healthy subjects: Healthy subjects with no known issues of increased gut permeability. These subjects will act as negative controls in all gut permeability studies.
  Interventions: Diagnostic Test: Spectroscopic gut permeability test
- 2b - Healthy subjects (gastric emptying): A subset of healthy volunteers will be recruited to take part in experiments to help in understanding the impact of gastric emptying rate as a confounding factor in measurements of gut permeability.
  Interventions: Diagnostic Test: Spectroscopic gut permeability test
- 3 - Increased permeability: Gastro-intestinal (GI) and non-GI patients who are expected to exhibit increased gut permeability (e.g. patients with celiac disease, inflammatory bowel disease (IBD), liver disease, HIV or another condition in which increased intestinal permeability is common). The more extreme cases in this group will act as positive controls.
  Interventions: Diagnostic Test: Spectroscopic gut permeability test

INTERVENTIONS:
Diagnostic Test: Spectroscopic gut permeability test — The spectroscopic gut permeability test first involves patients receiving an oral dose of one or more fluorescent dyes. A wearable sensor will then be attached to the patients' skin and this will be used to monitor the leakage of the fluorescent dyes from the intestine into the blood stream in a non-invasive manner. In this way, a measure of the permeability of the intestine will be obtained.
  Note that patients in Group 1 (ophthalmology patients) will not receive oral doses of contrast agents. Instead, the wearable sensor will simply be used to detect the presence of fluorescent dyes that were administered intravenously as part of planned ophthalmic procedures.
  Complete details of the spectroscopic gut permeability test can be found in the attached protocol.

SUMMARY:
This research aims to develop portable devices - known as fluorescence spectrometers - to monitor the leakage of fluorescent dyes out of the gut into the blood stream. These devices will measure the leakiness (permeability) of the gut in a non-invasive manner and will provide an early warning that patients are at risk of infections caused by the unwanted flow of bacteria from the intestine to the rest of the body.

DETAILED DESCRIPTION:
"Leaky gut" - or, increased permeability of the intestine - involves the leakage of certain intestinal constituents (e.g. endotoxins or even bacteria) from the gut into the rest of the body. This condition is associated with many widespread diseases including coeliac disease, inflammatory bowel disease, HIV, liver cirrhosis, sepsis and environmental enteric dysfunction (EED). It has a considerable impact on quality of life and, in extreme cases (e.g. sepsis), it can even lead to death. Furthermore, in the developing world (as part of EED), it severely hampers the mental and physical development of young children. Thus, new devices that can help us to learn more about leaky gut and more accurately monitor its effects are urgently needed.

In this project, patients will drink a small dose of a fluorescent dye. Then, by shining light on the patients' skin and recording the color and brightness of the light (fluorescence) that comes back, it will be possible to measure the amount of dye that has leaked into the blood (indicating the likelihood that bacteria are escaping from the gut and causing infections). We refer to this as a "Spectroscopic gut permeability test." We will also ask patients to take a traditional permeability test (known as a PEG permeability test) so that we can validate our new sensor. Overall, this research will deliver vital information that will improve our understanding of leaky gut and help guide the development of treatments for the many diseases in which it occurs.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Aged 18 years or above
* No evidence of prior adverse reactions to fluorescein, ICG, dextran or PEG
* No evidence of prior adverse reactions to iodine (for ICG experiments only)
* For healthy volunteers: healthy with no active GI/liver disease (or other condition in which increased gut permeability is expected, e.g. HIV) and no antibiotics taken within the previous four weeks.
* For cases: exhibiting symptoms of GI, liver or other diseases (e.g. HIV) in which increased intestinal permeability is expected.
* For ophthalmology patients recruited in Stage 1: healthy (i.e. as described above for healthy volunteers) and prescribed to have an ophthalmic angiography with an intravenous injection of either fluorescein or ICG.

Exclusion Criteria:

* Unable to give informed consent
* Aged <18 years
* Previous adverse reaction to fluorescein, ICG, dextran or PEG
* Known allergy to iodine (for ICG experiments only)
* Pregnancy (in Stage 1 this will be at the discretion of the patient's ophthalmologist)
* Breastfeeding (in Stage 1 this will be at the discretion of the ophthalmologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified and approached by members of their healthcare/clinical team. They will be identified based on their clinical condition and its potential relevance to the study - i.e. ophthalmology patients due to receive intravenous doses of fluorescein or ICG for Stage 1; GI and non-GI patients exhibiting increased intestinal permeability for Stages 2 and 3.
  Healthy volunteers with no indication of increased intestinal permeability will be recruited from Imperial College and St. Mary's Hospital staff. Potential healthy volunteers will be approached in person by members of the research team.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood concentration from intravenous injection | 1 day (study visit)
  Where the blood concentration of fluorescent dye is known - for example, in ophthalmology patients who have received a direct intravenous dose of contrast agent - a direct comparison will be made between these values and the results of the spectroscopic gut permeability test without the need for further measurements.
Blood concentration from samples | 1 day (study visit)
  In subjects receiving an oral dose of contrast agent, blood samples will be taken alongside the spectroscopic measurements in order to permit accurate ex vivo quantification of the serum concentration in the laboratory. These values will be compared with the spectroscopic findings.
PEG permeability assay | 1 week (after study visit)
  In patients who are also undergoing polyethylene glycol (PEG)-based permeability assays, spectroscopic permeability measurements will be compared to the results of this more traditional approach.
Histology | 1 day (study visit)
  Finally, in patients for whom intestinal biopsy and histology data is available, spectroscopic permeability measurements will be compared against histological measures of epithelial damage and permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Alex J Thompson, PhD, Principal Investigator — Imperial College London
Locations (1):
- IMPERIAL COLLEGE Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be made available to other researchers once the final results of the study have been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available once the final results of the study have been published. Data relevant to publications will be available indefinitely through a data repository. Additional data will be held on secure servers at Imperial College London for 10 years from the completion of the study.
Access Criteria: Data relevant to publications will be made available in an open access manner through data repositories. Additional data will be stored securely at Imperial College London for 10 years. Other researchers can request access to this data through the study chief investigator. This will be granted assuming that appropriate ethical approvals have been obtained.

REFERENCES:
- [Derived] Gan J, Chen Q, Monfort Sanchez E, Mandal N, Xu J, Wang Z, Agarwal A, Oluwatunmise E, Ramkumar P, Salam A, Chekmeneva E, Gomez-Romero M, Maslen L, Balarajah S, Perry R, Yong KK, Hoare J, Powell N, Alexander J, Avery J, Ashrafian H, Darzi A, Thompson AJ. Non-invasive fluorescence sensing reveals changes in intestinal barrier function and gastric emptying rate in a first-in-human study of Crohn's disease. Therap Adv Gastroenterol. 2025 Aug 13;18:17562848251361634. doi: 10.1177/17562848251361634. eCollection 2025. PMID 40821739

DOCUMENTS (5):
  • Informed Consent Form: ICF for ophthalmology patients (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT03434639/ICF_007.pdf
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03434639/Prot_SAP_008.pdf
  • Informed Consent Form: ICF for GI, liver and HIV patients (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03434639/ICF_009.pdf
  • Informed Consent Form: ICF for healthy volunteers (Group 2a) (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03434639/ICF_010.pdf
  • Informed Consent Form: ICF for healthy volunteers (Group 2b) (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT03434639/ICF_011.pdf